CLINICAL TRIAL: NCT01479296
Title: A Phase 1b Randomized Double-Blind Clinical Trial to Examine Whether Polytopic Administration of VRC rAd5 Gag-pol/Env A/B/C Vaccine Enhances HIV-Specific Cellular Immune Responses in Humans
Brief Title: Evaluating the Immune Response to a rAd5 HIV Vaccine Administered in Three Different Ways in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 085; 10796 (Other: DAIDS ES Registry Number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: rAd5 Plus Placebo (Experimental): Participants will receive the VRC rAd5 gag-pol/env A/B/C vaccine injection in their right arm (1×10^10 PU), and placebo vaccine injections in their left arm, right thigh, and left thigh.
  Interventions: Biological: VRC rAd5 vaccine (rAd5 gag-pol/env A/B/C); Biological: Placebo Vaccine
- Group 2: Separated Vaccine Components (Experimental): Participants will receive the rAd5 gag-pol vaccine injection in their right arm (0.5×10^10 PU), the rAd5 env A vaccine injection in their left arm (0.17×10^10 PU), the rAd5 env B vaccine injection in their right thigh (0.17×10^10 PU), and the rAd5 env C vaccine injection in their left thigh (0.17×10^10 PU).
  Interventions: Biological: rAd5 env A; Biological: rAd5 env B; Biological: rAd5 env C; Biological: rAd5 gag-pol
- Group 3: Divided Dose rAd5 (Experimental): Participants will receive the VRC rAd5 gag-pol/env A/B/C vaccine injection divided into fourths, with one fourth of the total dose given in each of 4 sites: right arm, left arm, right thigh, and left thigh (each at 0.25×10^10 PU).
  Interventions: Biological: VRC rAd5 vaccine (rAd5 gag-pol/env A/B/C)

INTERVENTIONS:
Biological: VRC rAd5 vaccine (rAd5 gag-pol/env A/B/C) — Given intramuscularly
  Other Names: VRC-HIVADV014-00-VP
  Arms: Group 1: rAd5 Plus Placebo; Group 3: Divided Dose rAd5
Biological: rAd5 env A — Given intramuscularly
  Other Names: VRC-HIVADV038-00-VP
  Arms: Group 2: Separated Vaccine Components
Biological: rAd5 env B — Given intramuscularly
  Other Names: VRC-HIVADV052-00-VP
  Arms: Group 2: Separated Vaccine Components
Biological: rAd5 env C — Given intramuscularly
  Other Names: VRC-HIVADV053-00-VP
  Arms: Group 2: Separated Vaccine Components
Biological: rAd5 gag-pol — Given intramuscularly
  Other Names: VRC-HIVADV054-00-VP
  Arms: Group 2: Separated Vaccine Components
Biological: Placebo Vaccine — Given intramuscularly
  Other Names: VRC-DILUENT013-DIL-VP
  Arms: Group 1: rAd5 Plus Placebo

SUMMARY:
The purpose of this study is to evaluate the immune response to the Vaccine Research Center (VRC) rAd5 HIV vaccine when the vaccine components are administered in three different ways, in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
The VRC rAd5 HIV vaccine contains four different components. In this study, researchers will examine how the immune system responds to the vaccine when the four components are administered in three different ways:

1. The vaccine dose containing all four components is given as a single injection in one arm, and placebo injections are given in the other arm and both legs.
2. The vaccine dose containing all four components is divided into fourths, and one-fourth of the full dose is given in each arm and leg.
3. The four vaccine components are separated, and a different component is given in each arm and leg.

This study will enroll healthy, HIV-uninfected adults. Participants will be randomly assigned to one of three groups. Group 1 will receive the entire dose of vaccine in their right arm and placebo vaccine in the other arm and both legs. Group 2 will receive all four different components of the vaccine, given separately as a different component per each arm and leg. Group 3 will receive the entire vaccine dose divided into fourths, with one fourth of the full dose given in each arm and leg.

At a baseline study visit, participants will undergo a physical examination and a medical and medication history review. Female participants will also take a pregnancy test. Participants will complete questionnaires and receive counseling on HIV risk reduction and pregnancy prevention. All participants will then receive vaccine given as four injections-one each in their right arm, left arm, right thigh, and left thigh (except for Group 1, placebo injections are given in left arm and both legs). After receiving the vaccine, participants will remain in the clinic for at least 30 minutes for observation and monitoring of side effects. For 7 days after the vaccination, participants will record any side effects in a symptom log; for the first 3 days after the vaccination, study staff will call participants to ensure they are completing the symptom log. Follow-up visits will occur at Months 1, 4, and 7. These visits will include the baseline study procedures and a blood collection. Participants will be contacted by study researchers once a year for 5 years for follow-up health monitoring. Blood collected during study visits will be saved for future testing.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willing to be followed for the planned duration of the study
* Able and willing to provide informed consent
* Demonstrates understanding of this study and that in a previous trial there was an association of increased acquisition of HIV with receipt of that study vaccine; completes a questionnaire prior to vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of exposure to HIV through the last required study visit
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 5 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required study visit (excludes annual contacts for safety surveillance)
* In good general health as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as being at "low risk" of HIV infection on the basis of sexual behaviors. More information on this criterion can be found in the protocol.
* Body weight greater than or equal to 110 lb (greater than or equal to 50 kg)
* Hemoglobin greater than or equal to 12.5 g/dL for participants who were born female; greater than or equal to 13.5 g/dL for participants who were born male
* White blood cell count between 3300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets between 125,000 to 550,000/mm^3
* Alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal
* Ad5 neutralizing antibody titer less than 1:18
* Negative HIV-1 and -2 blood test: U.S. participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA). Non-U.S. sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV) or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin pregnancy test performed prior to vaccination on the day of vaccination
* Participants who were born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through the last required study visit for sexual activity that could lead to pregnancy; or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation; or be sexually abstinent. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required study visit
* Participants who were born male must be fully circumcised (as documented at screening examination)

Exclusion Criteria:

* Excessive daily alcohol use, frequent binge drinking, chronic marijuana abuse, or any other use of illicit drugs within the 12 months prior to study entry
* History of newly acquired syphilis, gonorrhea, nongonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B within the 12 months prior to study entry
* Untreated or incompletely treated syphilis infection
* HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 085 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the 5 years prior to study entry in a previous vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For potential participants who have received control/placebo in an experimental vaccine trial, the HVTN 085 PSRT will determine eligibility on a case-by-case basis. For potential participants who have received an experimental vaccine(s) more than 5 years ago, eligibility for enrollment will be determined by the PSRT on a case-by-case basis.
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: 1) corticosteroid nasal spray for allergic rhinitis; 2) topical corticosteroids for mild, uncomplicated dermatitis; or 3) oral/parenteral corticosteroids given for nonchronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to study entry].)
* Blood products received within 120 days before the first vaccination
* Immunoglobulin received within 60 days before the first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before the first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to the first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before the first vaccination or that are scheduled within 14 days after the first vaccination
* Investigational research agents received within 30 days before the first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the study
* Current anti-tuberculosis prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, study adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy or thyroid disease requiring medication during the 12 months before study entry
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* Hypertension: If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at study entry or diastolic blood pressure greater than or equal to 100 mm Hg at study entry. More information on this criterion can be found in the protocol.
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with two or more of the following factors: age greater than or equal to 45 years old, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions)
* Cancer (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
* Seizure disorder (Not excluded: a participant with a history of seizures who has not required medications or had a seizure in the 3 years prior to study entry.)
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the study. Specifically excluded are people with psychoses within the 3 years prior to study entry, ongoing risk of suicide, or history of suicide attempt or gesture within the 3 years prior to study entry.
* Pregnant or breastfeeding
* Has been fully circumcised within 90 days prior to the first vaccination or displays evidence that surgical site is not fully healed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Number of recognized epitopes as measured by enzyme-linked immunospot (ELISpot) | Measured at 4 weeks following vaccination
Total magnitude of gene-specific CD4 and CD8 T-cell responses as measured by intracellular cytokine staining (ICS) | Measured at 4 weeks following vaccination

SECONDARY OUTCOMES:
Total vaccine-specific CD4 and CD8 T-cell responses as measured by ICS | Measured at 4 weeks following vaccination
Total vaccine-specific CD4 and CD8 T-cell responses as measured by ICS | Measured at 28 weeks following vaccination
Polyfunctional CD4 and CD8 T-cell responses across one and multiple antigenic components of VRC rAd5 HIV vaccine as measured by ICS | Measured at 28 weeks following vaccination
Antibody binding to HIV epitopes by multiplex binding antibody assay and/or peptide array | Measured at 28 weeks following vaccination
Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, adverse events (AEs), and serious adverse events (SAEs) reported on an expedited basis to the Division of AIDS (DAIDS) | Measured at 28 weeks following vaccination
T-cell receptor beta chain sequence diversity of epitope-specific CD4 and CD8 T cells | Measured at 28 weeks following vaccination
Human leukocyte antigen (HLA) type, epitope-specific T-cell responses as measured by ELISpot, ICS, tetramer, and/or other assays | Measured at 28 weeks following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ian Frank, Study Chair — University of Pennsylvania
Locations (8):
- United States (8):
  - Bridge HIV CRS, San Francisco, California
  - UIC Project WISH CRS, Chicago, Illinois
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

REFERENCES:
- [Background] Appay V, Douek DC, Price DA. CD8+ T cell efficacy in vaccination and disease. Nat Med. 2008 Jun;14(6):623-8. doi: 10.1038/nm.f.1774. PMID 18535580
- [Background] Vezys V, Yates A, Casey KA, Lanier G, Ahmed R, Antia R, Masopust D. Memory CD8 T-cell compartment grows in size with immunological experience. Nature. 2009 Jan 8;457(7226):196-9. doi: 10.1038/nature07486. Epub 2008 Nov 12. PMID 19005468